CLINICAL TRIAL: NCT07239804
Title: Systematic Assessment of Treatment Effectiveness for Long-Term Management of Stable Atrial Tachycardia in Inpatient and Outpatient Environments
Acronym: SATELLITE
Status: Active, not recruiting | Type: Observational
Sponsor: Evangelical Hospital Düsseldorf (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); Staedtisches Klinikum Karlsruhe (Other); Münster University Hospital, Germany (Unknown); Asklepios Klinik St. Georg (Unknown)
Responsible Party: Principal Investigator, Christian Meyer, Director of the Division of Cardiology, Electrophysiology, Angiology, Intensive Care at the EVK Düsseldorf and Principal Investigator, Evangelical Hospital Düsseldorf
Other Study IDs: SATELLITE
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Atrial Tachycardia; Stroke; Mortality; Atrial Flutter
Keywords: Atrial tachycardia rhythm control; Cardiovascular outcomes; Catheter ablation; Electrocardioversion; Stroke; Cardiac hospitalization; Mortality
MeSH Terms: conditions — Stroke; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing atrial tachycardia rhythm control: Patients undergoing catheter ablation and/or electrocardioversion for atrial tachycardia

SUMMARY:
The aim is to analyze long-term outcomes in a multicenter observational registry including patients undergoing atrial tachycardia rhythm control.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing atrial tachycardia rhythm control

Exclusion Criteria:

Follow-up <30 days after atrial tachycardia rhythm control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing atrial tachycardia rhythm control
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Mortality, stroke and cardiovascular hospitalization | From AT rhythm control through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, MD, MA, Principal Investigator — EVK, Düsseldorf
Locations (5):
- Germany (5):
  - EVK Düsseldorf, Düsseldorf
  - Asklepios Hospital St. Georg, Hamburg
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Municipal Clinical Center Karlsruhe, Karlsruhe
  - University Hospital Münster, Münster

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jungen C, Akbulak R, Kahle AK, Eickholt C, Schaeffer B, Scherschel K, Dinshaw L, Muenkler P, Schleberger R, Nies M, Gunawardene MA, Klatt N, Hartmann J, Merbold L, Jularic M, Willems S, Meyer C. Outcome after tailored catheter ablation of atrial tachycardia using ultra-high-density mapping. J Cardiovasc Electrophysiol. 2020 Oct;31(10):2645-2652. doi: 10.1111/jce.14703. Epub 2020 Aug 11. PMID 32748442
- [Background] Kahle AK, Jungen C, Scherschel K, Alken FA, Meyer C. Relationship Between Early and Late Recurrences After Catheter Ablation for Atrial Tachycardia in Patients With a History of Atrial Fibrillation. Circ Arrhythm Electrophysiol. 2022 Jun;15(6):e010727. doi: 10.1161/CIRCEP.121.010727. Epub 2022 May 27. No abstract available. PMID 35622433
- [Background] Brachmann J, Lewalter T, Kuck KH, Andresen D, Willems S, Spitzer SG, Straube F, Schumacher B, Eckardt L, Danilovic D, Thomas D, Hochadel M, Senges J. Long-term symptom improvement and patient satisfaction following catheter ablation of supraventricular tachycardia: insights from the German ablation registry. Eur Heart J. 2017 May 1;38(17):1317-1326. doi: 10.1093/eurheartj/ehx101. PMID 28329395